CLINICAL TRIAL: NCT03636477
Title: Protocol ATI001-102 Substudy: Evaluation of Ad-RTS-hIL-12 + Veledimex in Combination With Nivolumab in Subjects With Recurrent or Progressive Glioblastoma
Brief Title: A Study of Ad-RTS-hIL-12 With Veledimex in Combination With Nivolumab in Subjects With Glioblastoma; a Substudy to ATI001-102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI001-102 CPI Substudy 1.0
Record Dates: First submitted 2018-07-05; First posted 2018-08-17 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — veledimex; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ad-RTS-hIL-12 + veledimex in combination with nivolumab (Experimental): Intratumoral Ad-RTS-hIL-12 and varying doses of oral veledimex (activator ligand) given in combination with nivolumab via infusion.
  Interventions: Biological: Ad-RTS-hIL-12; Drug: veledimex; Drug: Nivolumab

INTERVENTIONS:
Biological: Ad-RTS-hIL-12 — * 2.0 x 10^11 viral particles (vp) per injection
  * intratumoral injection of Ad-RTS-hIL-12
Drug: veledimex — * 2 doses (10mg/day, 20mg/day)
  * 15 oral daily doses of veledimex
Drug: Nivolumab — * 2 doses (1mg/kg, 3mg/kg)
  * Every 2 weeks
  Other Names: Opdivo

SUMMARY:
This research study involves an investigational product: Ad-RTS-hIL-12 given with veledimex for production of human interleukin-12 (IL-12). IL-12 is a protein that can improve the body's natural response to disease by enhancing the ability of the immune system to kill tumor cells and may interfere with blood flow to the tumor.

Nivolumab is an antibody (a kind of human protein) that is being tested to see if it will allow the body's immune system to work against glioblastoma tumors. Opdivo (Nivolumab) is currently FDA approved in the United States for melanoma (a type of skin cancer), non-small cell lung cancer, renal cell cancer (a type of kidney cancer), Hodgkin's lymphoma but is not approved in glioblastoma. Nivolumab may help your immune system detect and attack cancer cells. Ad-RTS-hIL-12 and veledimex will be given in combination with Nivolumab to enhance the IL-12 mediated effect observed to date.

The main purpose of this substudy is to evaluate the safety and tolerability of a single tumoral injection of Ad-RTS-hIL-12 given with oral veledimex in combination with nivolumab.

DETAILED DESCRIPTION:
Eligible patients will receive one dose of nivolumab, via infusion, one week prior to standard of care craniotomy and tumor resection (subtotal or total). On the day of surgery, patients will receive one dose of veledimex before the resection procedure. Ad-RTS-hIL-12 will be administered by free-hand injection. Patients will continue on oral veledimex for 14 days. Following veledimex, patients will receive nivolumab via infusion every two weeks.

The study is divided into three periods: the screening period, the treatment period and the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥18 and ≤75 years of age
* Provision of written informed consent for tumor resection, stereotactic surgery, tumor biopsy, samples collection, and treatment with investigational products prior to undergoing any study specific procedures
* Histologically confirmed supratentorial glioblastoma
* Evidence of tumor recurrence/progression by magnetic resonance imaging (MRI) according to response assessment in neuro-oncology (RANO) criteria after standard initial therapy
* Previous standard-of-care antitumor treatment including surgery and/or biopsy and chemoradiation. At the time of registration, subjects must have recovered from the toxic effects of previous treatments as determined by the treating physician. The washout periods from prior therapies are intended as follows: (windows other than what is listed below should be allowed only after consultation with the Medical Monitor)

  1. Nitrosureas: 6 weeks
  2. Other cytotoxic agents: 4 weeks
  3. Antiangiogenic agents, including bevacizumab: 4weeks
  4. Targeted agents, including small molecule tyrosine kinase inhibitors: 2 weeks
  5. Vaccine-based therapy: 3 months
* Able to undergo standard MRI scans with contrast agent before enrollment and after treatment
* Karnofsky Performance Status ≥70%
* Adequate bone marrow reserves and liver and kidney function, as assessed by the following laboratory requirements:

  1. Hemoglobin ≥9 g/L
  2. Lymphocytes >500/mm3
  3. Absolute neutrophil count ≥1500/mm3
  4. Platelets ≥100,000/mm3
  5. Serum creatinine ≤1.5 x upper limit of normal (ULN)
  6. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 x ULN. For subjects with documented liver metastases, ALT and AST ≤5 x ULN
  7. Total bilirubin < 1.5 x ULN
  8. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) within normal institutional limits
* Male and female subjects must agree to use a highly reliable method of birth control (expected failure rate <5% per year) from the Screening Visit through 28 days after the last dose of study drug. Women of childbearing potential (perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential) must have a negative pregnancy test at screening.
* Normal cardiac and pulmonary function as evidenced by a normal electrocardiogram (ECG) and peripheral oxygen saturation (SpO2) ≥90% by pulse oximetry

Exclusion Criteria:

* Previous treatment with inhibitors of immunocheckpoint pathways (eg, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody) or other agents specifically targeting T cells
* Radiotherapy treatment within 4 weeks or less prior to veledimex dosing
* Subjects with clinically significant increased intracranial pressure (eg, impending herniation or requirement for immediate palliative treatment) or uncontrolled seizures
* Known immunosuppressive disease, or autoimmune conditions, and/or chronic viral infections (eg, human immunodeficiency virus [HIV], hepatitis)
* Use of systemic antibacterial, antifungal, or antiviral medications for the treatment of acute clinically significant infection within 2 weeks of first veledimex dose. Concomitant therapy for chronic infections is not allowed. Subjects must be afebrile prior to Ad-RTS-hIL-12 injection; only prophylactic antibiotic use is allowed perioperatively.
* Use of enzyme inducing antiepileptic drugs (EIAED) within 7 days prior to the first dose of study drug. Note: Levetiracetam (Keppra®) is not an EIAED and is allowed.
* Other concurrent clinically active malignant disease, requiring treatment, with the exception of non-melanoma cancers of the skin or carcinoma in situ of the cervix or nonmetastatic prostate cancer
* Nursing or pregnant females
* Prior exposure to veledimex
* Use of medications that induce, inhibit, or are substrates of cytochrome p450 (CYP450) 3A4 within 7 days prior to veledimex dosing without consultation with the Medical Monitor
* Presence of any contraindication for a neurosurgical procedure
* Unstable or clinically significant concurrent medical condition that would, in the opinion of the Investigator or Medical Monitor, jeopardize the safety of a subject and/or their compliance with the protocol. Examples include, but are not limited to: unstable angina, congestive heart failure, myocardial infarction within 2 months of screening, ongoing maintenance therapy for life-threatening ventricular arrhythmia or uncontrolled asthma.
* History of myocarditis or congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), as well as unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction 6 months prior to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaymes Holland, Study Director — Alaunos Therapeutics
Locations (4):
- United States (4):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Chiocca EA, Gelb AB, Chen CC, Rao G, Reardon DA, Wen PY, Bi WL, Peruzzi P, Amidei C, Triggs D, Seften L, Park G, Grant J, Truman K, Buck JY, Hadar N, Demars N, Miao J, Estupinan T, Loewy J, Chadha K, Tringali J, Cooper L, Lukas RV. Combined immunotherapy with controlled interleukin-12 gene therapy and immune checkpoint blockade in recurrent glioblastoma: An open-label, multi-institutional phase I trial. Neuro Oncol. 2022 Jun 1;24(6):951-963. doi: 10.1093/neuonc/noab271. PMID 34850166

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment and dose escalation followed a 3+3 design. Each subject in the 1st cohort, Cohort S1, was monitored through Day 28 before next subject was dosed. The first subjects in the subsequent cohorts, Cohorts S2 and S3, were monitored through Day 28. After completion of Cohort S3, the Safety Review Committee (SRC) and Data Safety Monitoring Board (DSMB )recommended expanding accrual, and additional 12 subjects were enrolled in an expansion cohort (20mg veledimex and 3mg/kg nivolumab).
Groups:
- Veledimex 10mg Dose Level + Nivolumab 1mg/kg: Cohort S1:
  Ad-RTS-hIL-12 on Day 0 Veledimex 10 mg once daily (QD) on Days 0-14 Nivolumab 1 mg/kg intravenously (IV) over 60 minutes on Day -7, Day 15, and approx every 2 weeks
- Veledimex 10mg Dose Level + Nivolumab 3mg/kg: Cohort S2:
  Ad-RTS-hIL-12 on Day 0 Veledimex 10 mg QD on Days 0-14 Nivolumab 3 mg/kg IV over 60 minutes on Day -7, Day 15, and approx every 2 weeks
- Veledimex 20mg Dose Level + Nivolumab 3mg/kg: Cohort S3:
  Ad-RTS-hIL-12 on Day 0 Veledimex 20 mg QD on Days 0-14 Nivolumab 3 mg/kg IV over 60 minutes on Day -7, Day 15, and approx every 2 weeks
Period: Overall Study
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Started | 3 | 3 | 15
Completed (Completed Veledimex treatment) | 3 | 3 | 14
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS): Overall Safety Population (OSP) includes all subjects who have received at least one dose of veledimex (pretumor resection and) and/or all subjects who received Ad-RTS-hIL-12.
Groups:
- Veledimex 10mg Dose Level + Nivolumab 1mg/kg: Cohort S1:
  Ad-RTS-hIL-12 on Day 0 Veledimex 10 mg QD on Days 0-14 Nivolumab 1 mg/kg IV over 60 minutes on Day -7, Day 15, and approx every 2 weeks
- Total: Total of all reporting groups
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 15 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 8 | 13
  >=65 years | 0 | 1 | 7 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.90 (17.34) | 59.37 (7.21) | 59.75 (13.54) | 57.29 (14.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 7 | 9
  Male | 2 | 2 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 14 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 14 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: cm] | 178.67 (8.93) | 175.27 (14.17) | 147.94 (10.15) | 175.52 (10.10)
Weight [Mean (Standard Deviation); unit: kg] | 74.33 (11.62) | 82.83 (29.11) | 85.19 (19.84) | 83.30 (19.71)
Disease Status at Entry [Count of Participants; unit: Participants]
  Unifocal | 2 | 3 | 10 | 15
  Multifocal | 1 | 0 | 5 | 6
  Missing | 0 | 0 | 0 | 0
Number of Recurrences [Count of Participants; unit: Participants]
  1st recurrence | 2 | 3 | 10 | 15
  >=2 recurrence | 1 | 0 | 4 | 5
  Missing | 0 | 0 | 1 | 1
Isocitrate Dehydrogenase (IDH) Mutation Status at Diagnosis [Count of Participants; unit: Participants] — Isocitrate Dehydrogenase: An enzyme involved in the citric acid cycle, crucial for cellular energy production. Mutations in the genes encoding this enzyme (IDH1 and IDH2) are associated with glioblastoma.
  Participants
    Mutated | 1 | 0 | 1 | 2
    Wild-Type | 2 | 3 | 14 | 19
    Missing | 0 | 0 | 0 | 0
MGMT Status at Diagnosis [Count of Participants; unit: Participants] — MGMT stands for O-6-methylguanine-DNA methyltransferase. It's a gene that makes a protein that helps repair damaged DNA in cells. Patients with methylated MGMT generally live longer, even without chemo. Patients with methylated MGMT respond better to temozolomide chemo.
  Participants
    Methylated | 2 | 1 | 5 | 8
    Unmethylated | 1 | 2 | 8 | 11
    Missing | 0 | 0 | 2 | 2
Karnofsky Performance Score (KPS) at Screening [Count of Participants; unit: Participants] — Karnofsky Performance Score is a way to measure how much a participant can do on their own.
  In this clinical trial, it was used to choose participants who were strong enough to handle treatment and give meaningful results. The score ranges from 100 to 0, in steps of 10:
  100 = Fully active, no symptoms. 70 = Able to care for self, but not do normal activities or work.
  Participants
    >= 70-90 | 0 | 0 | 4 | 4
    >= 90 | 3 | 3 | 11 | 17
    Missing | 0 | 0 | 0 | 0
Prior Lines of Treatment [Count of Participants; unit: Participants]
  Greater Than One | 0 | 0 | 5 | 5
  One | 3 | 3 | 10 | 16
Prior Steroid Use [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 3 | 3
  No | 3 | 3 | 12 | 18
  Missing | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Evaluation of adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.03 will be based on the incidence, intensity and type of adverse event.
  AEs will be regarded as treatment-emergent adverse events (TEAEs) during the treatment period regardless of relationship to study drug if:
  • The AE occurred or worsened from baseline during or after administration of the first dose of study drug (on or after Day 0).
Time Frame: 2 years and 4 months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 3 | 3 | 15
participants
  Any TEAEs | 3 | 3 | 15
  Any Serious TEAEs | 1 | 2 | 6
  Any TEAEs with Toxicity Grade ≥ 3 | 3 | 3 | 11
  Any TEAEs Leading to Treatment Dose Modification | 2 | 2 | 4
  Any TEAEs Leading to Treatment Discontinuations | 0 | 2 | 2
  Any TEAEs Leading to Death | 0 | 0 | 1
  Any Drug-Related TEAEs | 3 | 3 | 15
  Any Drug-Related Serious TEAEs | 1 | 1 | 3
  Any Drug-Related TEAEs with Toxicity Grade ≥ 3 | 2 | 3 | 7
  Any Drug-Related TEAEs Leading to Treatment Dose Modification | 2 | 1 | 4
  Any Drug-Related TEAEs Leading to Treatment Discontinuations | 0 | 1 | 2
  Any Drug-Related TEAEs Leading to Death | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Veledimex Dose Compliance
Description: Evaluation will be based on expected dose compliance. Subjects were instructed to document veledimex dosing compliance in a subject diary, including the time each dose was taken, the time of the last meal prior to administration of veledimex, the number of capsules taken, whether the subject missed any veledimex doses, and reason for any missed doses. Investigational product container(s) with any remaining capsules were returned to the study staff on Day 15, and staff assessed dose compliance.
Time Frame: From Day 0 through Day 14 for each participant
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 3 | 3 | 15
participants
  100% compliance | 2 | 3 | 11
  Less than 100% | 1 | 0 | 4
  80% or more | 3 | 3 | 15
  Less than 80% | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With a Dose-Limiting Toxicity (DLT)
Description: The primary objective was to determine the Maximum Tolerated Dose (MTD), defined as the dose at which fewer than 33% of subjects experience a Dose-Limiting Toxicity (DLT). The MTD was not reached; a Maximum Administered Dose (MAD) of 20mg veledimex and 3mg/kg nivolumab was determined. This measure reports the number of subjects who experienced a DLT during the first treatment cycle in each dose cohort.
Time Frame: The first treatment cycle (21 days).
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- Veledimex 10mg DoseLevel + Nivolumab1mg/kg: Cohort S1:
  Ad-RTS-hIL-12 on Day0 Veledimex 10 mg QD on Days 0-14 Nivolumab 1 mg/kg IV over 60 minutes on Day -7, Day 15, and approx every 2 weeks
- Veledimex 10mg Dose Level + Nivolumab 3mg/kg: Cohort S2:
  Ad-RTS-hIL-12 on Day0 Veledimex 10 mg QD on Days 0-14Nivolumab 3 mg/kg IV over 60 minutes on Day -7, Day 15, and approx every 2 weeks
- Veledimex 20mg Dose Level + Nivolumab 3mg/kg: Cohort S3:
  Ad-RTS-hIL-12 on Day0 Veledimex 20 mg QD on Days 0-14 Nivolumab 3 mg/kg IV over 60 minutes on Day -7, Day 15, and approx every 2 weeks
Arm/Group | Veledimex 10mg DoseLevel + Nivolumab1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 3 | 3 | 15
participants | 0 | 1 | 2

4. Secondary Outcome: Tumor Objective Response Rate (ORR)
Description: To determine investigator assessment of response including tumor ORR of Ad-RTS-hIL-12 + veledimex when administered in combination with nivolumab. Investigator assessment of ORR was determined according to Immunotherapy Response Assessment in Neuro-Oncology (iRANO) criteria. iRANO is a set of criteria built on RANO criteria but adapts them for immune-related effects to evaluate treatment response in brain tumor patients receiving immunotherapy. It addresses unique challenges like pseudoprogression, where immune-related inflammation mimics tumor growth on imaging allowing continued treatment despite early radiographic worsening if the patient is clinically stable. This criteria requires confirmation of progression with follow-up imaging ≥3 months later, especially within the first 6 months of immunotherapy.
Time Frame: 2 years and 4 months
Population: The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration. The ESP will be evaluated for investigator assessment of objective response rate (ORR).
Measure: Count of Participants; unit: Participants
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 3 | 3 | 15
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 1 | 0
  Stable Disease | 2 | 1 | 11
  Progressive Disease | 1 | 1 | 4
  Not Evaluable | 0 | 0 | 0
  No Response | 0 | 0 | 0
  Missing | 0 | 0 | 0

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is the time in days from the first treatment (either veledimex or Ad-RTS-hIL-12) to the first assessment on which the overall response is reported as disease progression (per Response Assessment in Neuro-Oncology [RANO] or Immunotherapy Response Assessment in Neuro-Oncology [iRANO] criteria). Subjects withdrawing from the study will be censored at their last non progressive disease response assessment. If a subject does not have a non-progressive disease response assessment, the subject will be censored on the date of the first treatment as described above.
Time Frame: 2 years and 4 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 3 | 3 | 15
Days | 38.0 (41.6) | 88.0 (98.8) | 36.9 (29.0)

6. Secondary Outcome: Rate of Pseudo-progression (PSP)
Description: PSP -- Progression free survival was originally defined for determination of PSP requiring confirmation of progression (per Response Assessment in Neuro-Oncology [RANO] or Immunotherapy Response Assessment in Neuro-Oncology [iRANO] criteria).
Time Frame: 2 years and 4 months
Population: The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration. The ESP is denoted as the PP population in this uncontrolled setting.
Measure: Number; unit: participants
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 3 | 3 | 15
participants | 0 | 1 | 0

7. Secondary Outcome: Overall Survival (OS)
Description: The percentage of participants alive at each time point (6, 9, 12, 15, 18, and 24 months) are reported.
Time Frame: Up to 24 months
Population: The Overall Safety Population (OSP) included all subjects who received at least one dose of any study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 3 | 3 | 15
Percentage of participants
  OS at Month 6 | 100 | 66.7 | 60.0
  OS at Month 9 | 66.7 | 66.7 | 46.7
  OS at Month 12 | 33.3 | 66.7 | 40
  OS at Month 15 | 33.3 | 66.7 | 26.7
  OS at Month 18 | 33.3 | 66.7 | 13.3
  OS at Month 24 | 0 | 33.3 | 0

8. Secondary Outcome: Changes From Baseline in Cellular Responses Elicited by Ad-RTS-hIL-12 and Veledimex in Combination With Nivolumab.
Description: Blood samples for pharmacodynamic biomarker evaluation were collected at screening, during treatment, and post-treatment. The immunological and biological response markers include serum cytokines (IL-12 and IFNℽ), and T and B cell subpopulations. Serum IL-12 and downstream IFNℽ expressions are reported by time point.
Time Frame: From Screening through Day 28, assessed at Screening and Days 0, 1, 3, 7, 14, and 28
Population: Evaluable Safety Population (ESP) includes subjects who have received nivolumab, Ad-RTS-hIL-12, and at least one dose of veledimex. Pharmacodynamic Population (PDP) refers to ESP.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 3 | 3 | 15
pg/mL
  Serum IL12 Screening: number analyzed (Participants) | 3 | 3 | 14
  Serum IL12 Screening | 1.19 (0.20) | 0.73 (0.15) | 0.40 (0.32)
  Serum IL12 Day 0 | 0.93 (0.26) | 1.12 (0.69) | 0.64 (0.34)
  Serum IL12 Day 1: number analyzed (Participants) | 3 | 3 | 14
  Serum IL12 Day 1 | 2.16 (2.03) | 0.90 (0.36) | 0.82 (0.38)
  Serum IL12 Day 3: number analyzed (Participants) | 3 | 3 | 14
  Serum IL12 Day 3 | 6.05 (3.70) | 2.22 (1.34) | 9.00 (11.57)
  Serum IL12 Day 7: number analyzed (Participants) | 1 | 2 | 11
  Serum IL12 Day 7 | 1.98 (0) | 3.84 (0.42) | 4.32 (3.82)
  Serum IL12 Day 14: number analyzed (Participants) | 2 | 3 | 14
  Serum IL12 Day 14 | 5.41 (4.75) | 1.01 (0.29) | 2.58 (2.49)
  Serum IL12 Day 28: number analyzed (Participants) | 3 | 3 | 13
  Serum IL12 Day 28 | 1.32 (0.50) | 0.84 (0.23) | 0.64 (0.33)
  Serum IFN gamma Screening | 8.93 (1.62) | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL. | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL.
  Serum IFN gamma Day 0 | 8.1 (0.17) | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL. | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL.
  Serum IFN gamma Day 1: number analyzed (Participants) | 3 | 3 | 14
  Serum IFN gamma Day 1 | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL. | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL. | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL.
  Serum IFN gamma Day 3: number analyzed (Participants) | 3 | 3 | 14
  Serum IFN gamma Day 3 | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL. | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL. | 2.12 (5.40)
  Serum IFN gamma Day 7: number analyzed (Participants) | 2 | 2 | 10
  Serum IFN gamma Day 7 | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL. | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL. | 5.46 (7.22)
  Serum IFN gamma Day 14: number analyzed (Participants) | 2 | 3 | 14
  Serum IFN gamma Day 14 | 13.9 (8.34) | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL. | 7.68 (28.73)
  Serum IFN gamma Day 28: number analyzed (Participants) | 3 | 3 | 13
  Serum IFN gamma Day 28 | NA (NA) — All values were below the limit of quantitation (BLQ) of 8 pg/mL. | 8.70 (1.21) | 3.52 (12.67)

9. Secondary Outcome: Changes From Baseline in Humoral Immune Responses Elicited by Ad-RTS-hIL-12 and Veledimex in Combination With Nivolumab.
Description: Blood samples for pharmacodynamic biomarker evaluation were collected at screening, during treatment, and post-treatment.
  Whole blood flow cytometry was used to assess the circulating blood cell subpopulations (e.g., T-reg and T cell panels).
Time Frame: From Screening through Day 28, assessed at Screening, Days 0, 14, and 28
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Combined: Veledimex 10mg Dose Level + Nivolumab 1mg/kg: Cohort S1:
  Ad-RTS-hIL-12 on Day 0 Veledimex 10 mg QD on Days 0-14 Nivolumab 1 mg/kg IV over 60 minutes on Day -7, Day 15, and approx every 2 weeks
Arm/Group | Combined: Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 3 | 3 | 15
percentage
  CD3+ CD45+ [pan-T] at Screening: number analyzed (Participants) | 2 | 2 | 14
  CD3+ CD45+ [pan-T] at Screening | 62 (15.56) | 78 (7.07) | 75 (14.14)
  CD3+ CD45+ [pan-T] at Day 0 | 58.67 (8.39) | 74.33 (7.51) | 75.5 (3.54)
  CD3+ CD45+ [pan-T] at Day 14 | 71.33 (7.37) | 73.67 (9.08) | 78 (3.83)
  CD3+ CD45+ [pan-T] at Day 28: number analyzed (Participants) | 3 | 3 | 14
  CD3+ CD45+ [pan-T] at Day 28 | 69 (7.55) | 77.33 (9.29) | 73 (2.83)
  CD3+ CD8+ [Tcytotoxic] at Screening: number analyzed (Participants) | 2 | 2 | 14
  CD3+ CD8+ [Tcytotoxic] at Screening | 21 (2.83) | 30.5 (0.71) | 32.5 (2.12)
  CD3+ CD8+ [Tcytotoxic] at Day 0 | 24 (3.61) | 31 (5) | 30 (4.24)
  CD3+ CD8+ [Tcytotoxic] at Day 14 | 31.67 (9.50) | 30.33 (1.15) | 29.5 (6.36)
  CD3+ CD8+ [Tcytotoxic] at Day 28: number analyzed (Participants) | 3 | 3 | 14
  CD3+ CD8+ [Tcytotoxic] at Day 28 | 29 (10.15) | 30.67 (4.62) | 31 (0)
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- [Treg] at Screening: number analyzed (Participants) | 2 | 2 | 13
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- [Treg] at Screening | 1.1 (0.57) | 1.8 (0.99) | 0.35 (0.49)
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- [Treg] at Day 0: number analyzed (Participants) | 3 | 2 | 12
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- [Treg] at Day 0 | 0.97 (0.38) | 0.85 (0.49) | 1.1 (0.99)
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- [Treg] at Day 14: number analyzed (Participants) | 3 | 3 | 13
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- [Treg] at Day 14 | 0.8 (0.78) | 1.70 (1.50) | 0.35 (0.35)
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- [Treg] at Day 28: number analyzed (Participants) | 3 | 2 | 13
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- [Treg] at Day 28 | 1.27 (1.24) | 2.9 (2.26) | 0.95 (0.92)

10. Secondary Outcome: Veledimex Pharmacokinetic Profile: Maximum Plasma Concentration (Cmax)
Description: Cmax was determined from the maximum plasma concentration from Day 0 (post veledimex and resection/craniotomy), 3-5 hours after the veledimex dose on Day 1, and 3-5 hours after the veledimex dose on Day 14.
Time Frame: Day 0 to Day 15 (Day 14 24-hour post dose)
Population: All subjects with available plasma-time concentration data are included in the PK Population.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Veledimex 10mg Dose Level + Nivolumab 1mg/kg: Cohort S1:
  Ad-RTS-hIL-12 on Day 0 Veledimex 10 mg QD on Days 0-14 Nivolumab 1 mg/kg IV over 60 minutes on Day -7, Day 15, and approx every 2 weeks
  Cohort S2:
  Ad-RTS-hIL-12 on Day 0 Veledimex 10 mg QD on Days 0-14 Nivolumab 3 mg/kg IV over 60 minutes on Day -7, Day 15, and approx every 2 weeks
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 2 | 3 | 15
ng/mL | 11.045 (6.159) | 13.707 (5.423) | 75.68 (82.38)

11. Secondary Outcome: Veledimex Pharmacokinetic Profile: Time to Maximum Plasma Concentration (Tmax)
Description: Tmax was determined from the time of maximum plasma concentration from Day 0 (post veledimex and resection/craniotomy), 3-5 hours after the veledimex dose on Day 1, and 3-5 hours after the veledimex dose on Day 14.
Time Frame: Day 0 to Day 15 (Day 14 24-hour post dose)
Population: All subjects with available plasma-time concentration data are included in the PK Population.
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Combined: Veledimex 10mg Dose Level + Nivolumab 1mg/kg & 3mg/kg: Cohort S1:
  Ad-RTS-hIL-12 on Day 0 Veledimex 10 mg QD on Days 0-14 Nivolumab 1 mg/kg IV over 60 minutes on Day -7, Day 15, and approx every 2 weeks
Arm/Group | Combined: Veledimex 10mg Dose Level + Nivolumab 1mg/kg & 3mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 2 | 3 | 15
Hours | 3.95 (0.12) | 4.00 (1.18) | 4.63 (2.79)

12. Secondary Outcome: Veledimex Pharmacokinetic Profile: Half-life (t1/2)
Description: t1/2 was determined from the plasma concentrations measured from Day 0 (post veledimex and resection/craniotomy) through Day 15 (24 hours post Day 14 dose)
Time Frame: Day 0 to Day 15 (24 hours post Day 14 dose)
Population: All subjects with available plasma-time concentration data are included in the PK Population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 2 | 3 | 15
hours | 1.39 (0.14) | 1.79 (0.50) | 1.63 (0.77)

13. Secondary Outcome: Veledimex Pharmacokinetic Profile: Area Under the Concentration-versus-time Curve (AUC)
Description: AUC was determined from the plasma concentrations measured from Day 0 (post veledimex and resection/craniotomy) through Day 15 (24 hours post Day 14 dose)
Time Frame: Day 0 to Day 15 (Day 14 24-hour post dose)
Population: All Subjects with available plasma-time concentration data are included in the PK Population.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 2 | 3 | 15
ng*hr/mL | 24.85 (13.82) | 30.76 (5.42) | 185.34 (215.77)

14. Secondary Outcome: Veledimex Pharmacokinetic Profile: Volume of Distribution (Vd)
Description: Vd was determined from the plasma concentrations measured from Day 0 (post veledimex and resection/craniotomy) through Day 15 (24 hours post Day 14 dose).
Time Frame: Day 0 to Day 15 (Day 14 24-hour post dose)
Population: All subjects with available plasma-time concentration data are included in the PK Population.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 2 | 3 | 15
L | 1.07 (0.60) | 0.83 (0.39) | 0.53 (0.37)

15. Secondary Outcome: Veledimex Pharmacokinetic Profile: Clearance (CL)
Description: CL was determined from the plasma concentrations measured from Day 0 (post veledimex and resection/craniotomy) through Day 15 (24 hours post Day 14 dose).
Time Frame: Day 0 to Day 15 (Day 14 24-hour post dose)
Population: All subjects with available plasma-time concentration data are included in the PK Population.
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 2 | 3 | 15
L/hour | 0.476 (0.265) | 0.332 (0.060) | 0.219 (0.142)

16. Secondary Outcome: Veledimex Concentration Ratio Between the Brain Tumor and the Blood.
Description: Tumor/plasma ratio at Day 0 by cohort
Time Frame: 1 day (Day 0 at time of resection)
Population: All subjects with available tumor concentration data are included in the PK Population for determination of tumor/plasma concentration ratio.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 3 | 2 | 14
ratio | 0.561 (0.212) | 0.404 (0.87) | 0.632 (0.446)

17. Secondary Outcome: Cumulative Dexamethasone Use During Days 0-14
Description: To assess concomitant corticosteroid use during the first treatment cycle, the cumulative dose of dexamethasone administered to each subject from Day 0 to Day 14 was calculated. This measure reports the mean cumulative dose in milligrams (mg) for each cohort
Time Frame: Days 0 through 14
Population: The Overall Safety Population (OSP) includes all subjects who have received at least one dose of veledimex and/or Ad-RTS-hIL-12
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
Number analyzed (Participants) | 3 | 3 | 15
mg | 82.7 (88.6) | 20 (0) | 60.1 (100.2)

ADVERSE EVENTS:
Time Frame: 2 years and 4 months
Description: The Full Analysis Set (FAS): Overall Safety Population (OSP) includes all subjects who have received at least one dose of veledimex (pretumor resection and) and/or all subjects who received Ad-RTS-hIL-12.
  AEs will be regarded as treatment-emergent TEAEs during the treatment period regardless of relationship to study drug if:
  • The AE occurred or worsened from baseline during or after administration of the first dose of study drug (on or after Day 0).
Arm/Group | Veledimex 10mg Dose Level + Nivolumab 1mg/kg | Veledimex 10mg Dose Level + Nivolumab 3mg/kg | Veledimex 20mg Dose Level + Nivolumab 3mg/kg
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 15/15
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 6/15
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veledimex 10mg Dose Level + Nivolumab 1mg/kg (N=3) | Veledimex 10mg Dose Level + Nivolumab 3mg/kg (N=3) | Veledimex 20mg Dose Level + Nivolumab 3mg/kg (N=15)
Brain Oedema (Nervous system disorders) | 1 (1) | 1 (2) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cold Type Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cytokine Release Syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Immune Reconstitution Inflammatory Syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veledimex 10mg Dose Level + Nivolumab 1mg/kg (N=3) | Veledimex 10mg Dose Level + Nivolumab 3mg/kg (N=3) | Veledimex 20mg Dose Level + Nivolumab 3mg/kg (N=15)
Headache (Nervous system disorders) | 2 (3) | 3 (4) | 13 (15)
Seizure (Nervous system disorders) | 1 (2) | 0 (0) | 3 (7)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1) | 5 (10)
Aphasia (Nervous system disorders) | 1 (2) | 2 (2) | 2 (4)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Facial Paresis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Hemianopia Homonymous (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Neurologic Neglect Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Visual Field Defect (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Apraxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrospinal Fluid Leakage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Quadrantanopia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 2 (4) | 2 (2) | 9 (20)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 2 (6) | 5 (10)
Alanine Aminotransferase Increased (Investigations) | 1 (3) | 0 (0) | 4 (5)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 4 (5)
Lipase Increased (Investigations) | 0 (0) | 1 (3) | 2 (2)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 3 (4)
Neutrophil Count Decreased (Investigations) | 0 (0) | 1 (3) | 2 (3)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Amylase Increased (Investigations) | 0 (0) | 1 (4) | 1 (2)
Body Temperature Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
International Normalised Ratio Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 8 (8)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 5 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (8) | 5 (11)
Fatigue (General disorders) | 1 (1) | 1 (1) | 4 (4)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (5) | 6 (9)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Flat Affect (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Personality Change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Procedural Headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Urethral Pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Cytokine Release Syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Brain Oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure shall not occur until (i) twenty-four (24) months have elapsed since Sponsor has notified Institution of the completion of the multi-center Study in order for Sponsor to comply with its obligations under 21 CFR 312.53(c)(4), or (ii) after the publication of the multi-center Study data, if the Study is a multi-center Study or Sponsor confirms in writing there will be no multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT03636477/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT03636477/SAP_001.pdf